CLINICAL TRIAL: NCT00288379
Title: A Comparative, Placebo-controlled, Double Blind, Double Dummy, Cross-over, Single Centre, Phase IIIb Study Between Formoterol Alone (Oxis® Turbuhaler® 4.5 µg) and the Fixed Combination of Formoterol and Budesonide (Symbicort® Turbuhaler®160/4.5 µg) on Airway Responsiveness and Airway Inflammation Induced by Repeated Low-dose Allergen Challenge in Allergic Patients With Mild Asthma
Brief Title: SMILDA - Symbicort®Turbuhaler® Allergan Challenge Study in Allergic Patients With Mild Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D5890L00007; EudraCT No 2004-000211-26
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma; allergen challenge; airway responsiveness; airway inflammation; Symbicort®
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

INTERVENTIONS:
Drug: formoterol
Drug: budesonide/formoterol

SUMMARY:
To compare the effects of formoterol alone (Oxis® TurbuhalerÒ) and the fixed combination of formoterol and budesonide (Symbicort® TurbuhalerÒ) on airway responsiveness as a marker of inflammation, induced by repeated low-dose allergen challenge in allergic patients with mild asthma

ELIGIBILITY:
Inclusion Criteria:

* A diagnosed history of asthma for at least 6 months
* Mild and stable asthma, only using β2-agonists as needed for the last 4 weeks.
* FEV1 >70% of predicted normal value (post-bronchodilator value).
* Skin prick test positive to pollen, animal dander or house dust mite.

Exclusion Criteria:

* Any significant respiratory disease, other than asthma.
* Upper or lower respiratory tract infection within 4 weeks before inclusion.
* Use of:

  1. inhaled glucocorticosteroid treatment for the last 8 weeks prior to inclusion or ever used oral glucocorticoid treatment for asthma.
  2. inhaled long-acting or oral b2-agonists, anticholinergic bronchodilators, cromones, antihistamines, theophyllines and anti-leukotrienes within 2 weeks of screening.
  3. regular NSAIDs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16
Dates: Start 2004-10; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
PD20 methacholine (measured as the change using the measurement before and after each treatment period).

SECONDARY OUTCOMES:
eNO (ppb).
Forced Expiratory Volume in one second (FEV1 ) - Induced sputum:
Total and differential blood cell count
Different Biomarkers
Safety endpoints will be incidence of Serious Adverse Events (SAEs)
Discontinuation due to Adverse Events (DAEs).

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Symbicort Medical Science Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Stockholm, Sweden